CLINICAL TRIAL: NCT06174454
Title: Clinical Efficacy of Respiratory Pediatric Physiotherapy on a Child With Hospital Treated Pneumonia: Single-Blind Clinical Trial
Brief Title: Clinical Efficacy of Respiratory Pediatric Physiotherapy on a Child With Hospital Treated Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Adrian Morales Muñoz, Principal Investigator, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HIM2017-055 SSA1376
Record Dates: First submitted 2018-02-18; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Pneumonia Childhood; Rehabilitation; Recovery of Function
Keywords: Pneumonia; Respiratory Pediatric Physiotherapy
MeSH Terms: conditions — Pneumonia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The population will consist of children aged from 0 to 8 years old diagnosed with pneumonia with a development time less than 7 days. he sample calculation corresponds to 40 participants per group. The intervention group will be exposed to techniques such as prolonged slow expiration, controlled expiratory flow exercises, tracheal pumping and tracheal reflex. The control group will be subject to postural drainage plus compressions to the muscle belly of the upper limbs. Both groups will go through 10 sessions: One daily session from Monday to Friday with a duration of 10 to 15 minutes each
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: 1. A sequence of aleatory numbers in blocks of 2 will be generated in each of the study groups using the software randomization.com, done by a person foreign to the research.
  2. Using the randomized numbers generated by the software, it will be decided what group each participant belongs to (control or intervention) and what maneuver will be assigned to them.
  3. These numbers and their maneuvers will be placed inside dark envelopes.
  4. The whole randomization and assignment sequence will be performed by a person foreign to the research and without the knowledge of the researchers. Support will be provided from the coordination for nursing research, who will select the personnel for the process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inervention group (Experimental): The intervention group will be subject to RPP. Techniques of slow expiration will be used and slow inspiration for the sweeping of secretions, during its expulsion forced expiratory techniques will be used (tracheal reflex). 10 sessions will be performed, one a day from Monday to Friday, with a duration of 10 to 15 minutes.
  Interventions: Other: Respiratory Pediatric Physiotherapy
- Control Group (Placebo Comparator): Will be subject to PD plus muscle belly compressions of the upper limbs for 10 sessions, one session a day from Monday to Friday, with a duration de 10 to 15 minutes per patient. Both groups will receive the usual treatment for pneumonia prescribed by their treating doctor.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Respiratory Pediatric Physiotherapy — Prolonged slow expiration Tracheal pumping Controlled expiratory flow exercises Forced expiration technique
  Other Names: Fisioterapia torácica pediatrica
  Arms: Inervention group
Other: Control Group — Will be subject to muscle compressions of the upper limbs. Both groups will receive the usual treatment for pneumonia prescribed by their treating doctor.
  Arms: Control Group

SUMMARY:
The accumulation of secretions in the bronchopulmonary air network promotes the detriment of respiratory functions generating hypoxia and causing a decrease in the cardiac output requiring the use of mechanical ventilation and hemodynamic support. It is intended to control the accumulation of secretions by means of Respiratory Pediatric Physiotherapy (RPP) and to evaluate its effectiveness counting on biological plausibility.

DETAILED DESCRIPTION:
The OBJECTIVE of this research protocol is to evaluate the effectiveness of RPP compared to postural drainage plus compression to the muscle belly of the upper limbs, as an adjuvant treatment for children with pneumonia. It is expected that the clinical severity decreases by 1.5 in the Wang score (a modification of the Silverman score), with a standard deviation of 2.6 points and a decrease of two days in the hospital stay with a α 0.05 in a one-tail test, a P of 80% and a 95.5% confidence interval.

ELIGIBILITY:
Inclusion criteria:

1. Patients from the Hospital Infantil de México Federico Góme with diagnosis of pneumonia (considering the diagnostic criteria of the WHO and the Guidelines for Nosocomial Pneumonia from the infectiology department.
2. Patients aged 0 to 8 years old.
3. A minimum HS of 72 hours.
4. Having informed consent.
5. Not having had previous RPP treatment.

Exclusion Criteria:

1. Presenting a fever state for more than three days. Performing physiotherapy increases the body's peripheral temperature.
2. Presenting an oxygen saturation below 80%.
3. Requiring mechanical ventilation.
4. Hemodynamic instability.
5. Presenting systemic inflammatory response syndrome.
6. Inotropic support.
7. Anatomical variants in the thorax.
8. Unstable thorax.
9. Esophageal atresia.
10. Pleural effusion, pneumothorax.
11. Alterations that compromise respiratory centers and/or the phrenic nerve.
12. Neuromuscular diseases that compromise respiratory mechanics.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2018-02-03 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-11-04 (Actual)

PRIMARY OUTCOMES:
Respiratory difficulty | 5 days
  The Silverman score will be used with a range of 0 to 10 points, directly proportional between the sum and the respiratory difficulty.

SECONDARY OUTCOMES:
Hospital stay | 7 days
  Days of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Morales, Fisioterapia, Principal Investigator — Hospital Infantil de Mexico Federico Gomez
Locations (1):
- Hospital Infantil de México Federico Gómez, Mexico City, Delegación Cuauhtémoc, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Girardi G, et al. El Programa IRA en Chile: hitos e historia. Chil Ped (Chil). 2001; 72: 292-300.
- [Background] European Respiratory Society Annual Congress. Effects of a new chest physiotherapy protocol in infant RSV bronchiolitis; 4-8 october. Berlín: European Respiratory Society; 2008.
- [Result] Postiaux G, Hankard R, Saulnier JP, Karolewicz S, Benielli J, Le Dinahet T, Louis J. Chest physical therapy in infant acute viral bronchiolitis: should we really surrender? Arch Pediatr. 2014 May;21(5):452-3. doi: 10.1016/j.arcped.2014.02.029. Epub 2014 Apr 8. No abstract available. PMID 24721416

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT06174454/Prot_SAP_000.pdf